CLINICAL TRIAL: NCT00893854
Title: The Comparison Between the Therapeutic Affect of Intravitreal Diclophenac and Triamcinolone in Persistent Uveitic Cystoids Macular Edema
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8727
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-05

CONDITIONS: Uveitis; Cystoid Macular Edema
MeSH Terms: conditions — Uveitis; Macular Edema | interventions — Diclofenac; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclophenac (Experimental)
  Interventions: Drug: Diclophenac
- Triamcinolone (Experimental)
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: Diclophenac
  Arms: Diclophenac
Drug: Triamcinolone
  Arms: Triamcinolone

SUMMARY:
Cystoids macular edema (CME) is one of the most common causes of low vision due to uveitis. The treatment for reducing the intra-ocular inflammation can decrease the macular edema. In some patients, CME persists even after inflammation control, and additional treatment is needed for better vision. Oral steroid, periocular and intravitreal Triamcinolone are the principles in treatment, but some complications like cataracts and increased ocular pressure have been seen. Diclophenac is a non-steroid anti-inflammatory drug that improves the vision and decreases the macular thickness by slowing down the prostaglandin E2 (PGE2) ending in vascular endothelial growth factor (VEGF) inhibition. In this study, the investigators are going to compare the therapeutic affect of intravitreal Diclophenac and Triamcinolone in persistent uveitic cystoids macular edema. Since diclophenac is a cheap and accessible drug in all curative centers it could be applied instead of Triamcinolone.

ELIGIBILITY:
Inclusion Criteria:

* cystoids macular edema which is diagnosed by OCT and flurocein angiography
* 5/200 < Visual acuity < 20/50
* resistance to routine treatment (oral treatment, periocular injection)

Exclusion Criteria:

* history of retinal disease cause macular edema like diabetes
* arterial occlusion
* monocular patients
* patients candidate for intra-ocular operation
* history of glaucoma or ocular hypertension
* any cataract that would interfere with OCT

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran